CLINICAL TRIAL: NCT03812770
Title: Sorafenib Plus Hepatic Artery Infusion Chemotherapy of Oxaliplatin, Fluorouracil/Leucovorin Versus Sorafenib Plus Hepatic Artery Infusion Chemotherapy of Oxaliplatin for Advanced Hepatocellular Carcinoma
Brief Title: Phase 2 Study of Sorafenib Plus HAIC of FOLFOX vs. Sorafenib Plus HAIC of OXA for Advanced HCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Kaiping Central Hospital (Other); Guangzhou No.12 People's Hospital (Other Government)
Responsible Party: Principal Investigator, Shi Ming, Clinical Professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC-OXA
Record Dates: First submitted 2019-01-19; First posted 2019-01-23 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Sorafenib; Hepatic artery infusion chemotherapy; Oxaliplatin, 5-Fluorouracil and Leucovorin; Oxaliplatin
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib; Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sorafenib plus HAIC of OXA (Experimental): Sorafenib combined with Hepatic arterial infusion chemotherapy with Oxaliplatin
  Interventions: Drug: Sorafenib; Drug: HAIC of OXA
- Sorafenib plus HAIC of FOLFOX (Active Comparator): Sorafenib combined with Hepatic arterial infusion chemotherapy with Oxaliplatin, Fluorouracil and Leucovorin
  Interventions: Drug: Sorafenib; Drug: HAIC of FOLFOX

INTERVENTIONS:
Drug: Sorafenib — Oral Sorafenib, 400mg, Bid
Drug: HAIC of FOLFOX — administration of Oxaliplatin , fluorouracil, and leucovorin via the tumor feeding arteries
  Other Names: Oxaliplatin , fluorouracil, and leucovorin
  Arms: Sorafenib plus HAIC of FOLFOX
Drug: HAIC of OXA — administration of Oxaliplatin via the tumor feeding arteries
  Other Names: Oxaliplatin
  Arms: Sorafenib plus HAIC of OXA

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of hepatic arterial infusion chemotherapy (HAIC) of oxaliplatin plus fluorouracil/leucovorin compared with HAIC of oxaliplatin alone in patients with advanced hepatocellular carcinoma (HCC)

DETAILED DESCRIPTION:
Sorafenib is the most widely used palliative treatment for advanced hepatocellular carcinoma (HCC) patients . Our previous prospective study revealed that sorafenib combined with hepatic arterial infusion chemotherapy (HAIC) of oxaliplatin plus fluorouracil/leucovorin confer a survival benefit to advanced HCC . However, HAIC of fluorouracil is not such for advanced HCC. Whether HAIC of oxaliplatin is as effective as HAIC of oxaliplatin plus fluorouracil/leucovorin is controversial. Thus, the investigators carried out this prospective randomized control study to find out it.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of HCC was based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL)
* Patients must have at least one tumor lesion that can be accurately measured according to EASL criteria.
* Barcelona clinic liver cancer-stage C
* Eastern Cooperative Oncology Group performance status of 0 to 2
* with no previous treatment
* No Cirrhosis or cirrhotic status of Child-Pugh class A only
* Not amendable to surgical resection ,local ablative therapy and any other cured treatment.
* The following laboratory parameters:

Platelet count ≥ 75,000/μL Hemoglobin ≥ 8.5 g/dL Total bilirubin ≤ 30mmol/L Serum albumin ≥ 30 g/L ASL and AST ≤ 5 x upper limit of normal Serum creatinine ≤ 1.5 x upper limit of normal INR ≤ 1.5 or PT/APTT within normal limits Absolute neutrophil count (ANC) >1,500/mm3

• Ability to understand the protocol and to agree to and sign a written informed consent document

Exclusion Criteria:

* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of bleeding diathesis.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug
* Serious non-healing wound, ulcer, or bone fracture
* Known central nervous system tumors including metastatic brain disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-08-04 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 12 months
  PFS was defined as the time from the date of randomization to the date of first documentation of disease progression based on modified Response Evaluation Criteria in Solid Tumors (mRECIST), or date of death, whichever occurred first.

SECONDARY OUTCOMES:
Overall Survival (OS) | 12 months
  OS was defined as the duration from the date of randomization until the date of death from any cause. Participants who were lost to follow-up were censored at the last date the participant was known to be alive, and participants who remained alive were censored at the time of data cutoff.
Objective Response Rate (ORR) | 12 months
  ORR was defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR) based on mRECIST. CR was defined as disappearance of any intratumoral arterial enhancement in all target lesions. PR was defined as at least a 30% decrease in the sum of diameters of viable (enhancement of arterial phase) target lesions taking as reference to the baseline sum of the diameters of target lesions.
Adverse Events | 30 days
  Number of adverse events. Postoperative adverse events were graded based on CTCAE v4.03

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Cancer Center Sun Yat-sen University, Guangzhou, Guangdong
  - Guangzhou Twelfth People 's Hospita, Guangzhou, Guangdong
  - Kaiping Central Hospital, Kaiping, Guangdong